CLINICAL TRIAL: NCT01060072
Title: A Randomized, Multicenter, Double-Masked, Parallel-Group Clinical Safety and Efficacy Evaluation of Loteprednol Etabonate, 0.5% Versus Vehicle for the Treatment of Inflammation and Pain Following Cataract Surgery
Brief Title: Evaluation of Loteprednol Etabonate Versus Vehicle for the Treatment of Inflammation and Pain Following Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 577
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Results first posted 2012-01-13 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2011-12

CONDITIONS: Inflammation; Pain
MeSH Terms: conditions — Inflammation; Pain | interventions — Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loteprednol etabonate (Experimental): Loteprednol etabonate 0.5% ophthalmic suspension
  Interventions: Drug: Loteprednol etabonate
- Vehicle (Placebo Comparator): Vehicle of loteprednol etabonate ophthalmic suspension
  Interventions: Drug: Vehicle of Loteprednol Etabonate

INTERVENTIONS:
Drug: Loteprednol etabonate — Topical administration of loteprednol etabonate ophthalmic suspension 1-2 drops in study eye four times a day (QID), postoperative day 1-14.
  Arms: Loteprednol etabonate
Drug: Vehicle of Loteprednol Etabonate — Topical administration of vehicle of loteprednol etabonate ophthalmic suspension 1-2 drops in study eye QID, postoperative day 1-14.
  Arms: Vehicle

SUMMARY:
This study is being conducted to compare the safety and efficacy of loteprednol etabonate to vehicle for the treatment of postoperative inflammation and pain following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are at least 18 years of age.
* Subjects who are candidates for routine, uncomplicated cataract surgery.

Exclusion Criteria:

* Subjects who have known hypersensitivity or contraindication to the study drug or components.
* Subjects with a severe/serious ocular condition, or any other unstable medical condition, that in the investigator's opinion may preclude study treatment or follow-up.
* Subjects with elevated intraocular pressure (>/=21mm Hg), uncontrolled glaucoma, or being treated for glaucoma in the study eye.
* Subjects who are monocular or have pinholed Snellen visual acuity (VA) 20/200 or worse in the non-study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2010-02; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Trusso, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Rochester, New York, United States

REFERENCES:
- [Derived] Rajpal RK, Fong R, Comstock TL. Loteprednol etabonate ophthalmic gel 0.5% following cataract surgery: integrated analysis of two clinical studies. Adv Ther. 2013 Oct;30(10):907-23. doi: 10.1007/s12325-013-0059-7. Epub 2013 Oct 18. PMID 24136301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 22 enrolling sites; 2 in the European Union (EU) and 20 in the United States (US). First participant was enrolled on 2/19/2010 and last participant completed the study on 9/3/2010.
Pre-assignment Details: A total of 407 participants, who were candidates for routine, uncomplicated cataract surgery, were enrolled in the study, 400 participants completed the study.
Period: Overall Study
Arm/Group | Loteprednol Etabonate | Vehicle
Started | 206 | 201
Completed | 204 | 196
Not Completed | 2 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Acute cholecystitis | 1 | 0
Not completed — Excluded Medications | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loteprednol Etabonate | Vehicle | Total
Number analyzed (Participants) | 206 | 201 | 407
Age Continuous [Mean (Standard Deviation); unit: years] — Intent to treat Population (ITT)
  years | 68.3 (9.66) | 69.4 (9.56) | 68.9 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 109 | 233
  Male | 82 | 92 | 174
Region of Enrollment [Number; unit: participants]
  United States | 198 | 193 | 391
  Germany | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Resolution of Anterior Chamber Cells.
Description: Participants with complete resolution of anterior chamber cells(ACC). Cells were graded on a 0-4 scale, where 0=no cells and 4=>30 cells
Time Frame: Visit 5 (Postoperative day 8)
Population: Intention to treat (ITT) population
Measure: Number; unit: participants
Arm/Group | Loteprednol Etabonate | Vehicle
Number analyzed (Participants) | 206 | 201
participants | 64 | 28

2. Primary Outcome: Grade 0 Pain
Description: Participants with no pain, graded on a 0-5 scale, 0=no pain and 5=severe pain
Time Frame: Visit 5 (Postoperative day 8)
Population: Intention to treat (ITT) population
Measure: Number; unit: participants
Arm/Group | Loteprednol Etabonate | Vehicle
Number analyzed (Participants) | 206 | 201
participants | 156 | 92

3. Secondary Outcome: Resolution of Anterior Chamber Cells
Description: as for outcome 1
Time Frame: Visit 4-7 (postoperative day 3-18)
Population: Intention to treat population (ITT)
Measure: Number; unit: participants
Arm/Group | Loteprednol Etabonate | Vehicle
Number analyzed (Participants) | 206 | 201
participants
  Visit 4 (Postoperative Day 3) | 8 | 7
  Visit 5 (Postoperative Day 8) | 64 | 28
  Visit 6 (Postoperative Day 15) | 116 | 61
  Visit 7 (Postoperative Day 18) | 114 | 59

4. Secondary Outcome: Grade 0 Pain
Description: Participants with no pain, graded on a 0-5 scale, 0= no pain and 5=severe pain
Time Frame: Visits 4-7 (Postoperative days 3-18)
Population: Intention to treat population (ITT)
Measure: Number; unit: participants
Arm/Group | Loteprednol Etabonate | Vehicle
Number analyzed (Participants) | 206 | 201
participants
  Visit 4 (Postoperative Day 3) | 139 | 93
  Visit 5 (Postoperative Day 8) | 156 | 92
  Visit 6 (Postoperative Day 15) | 160 | 89
  Visit 7 (Postoperative Day 18) | 151 | 79

5. Secondary Outcome: Resolution of Anterior Chamber Flare
Description: Complete resolution of flare, scored on a scale of 0-4 were 0=none and 4=very severe.
Time Frame: Visit 4-7 (postoperative day 3-18)
Population: Intention to treat population (ITT)
Measure: Number; unit: participants
Arm/Group | Loteprednol Etabonate | Vehicle
Number analyzed (Participants) | 206 | 201
participants
  Visit 4 (Postoperative Day 3) | 93 | 64
  Visit 5 (Postoperative Day 8) | 134 | 72
  Visit 6 (Postoperative Day 15) | 162 | 90
  Visit 7 (Postoperative Day 18) | 143 | 75

ADVERSE EVENTS:
Time Frame: 14 Days
Arm/Group | Loteprednol Etabonate | Vehicle
Serious Adverse Events (participants affected / at risk) | 3/206 | 1/201
Other Adverse Events (participants affected / at risk) | 10/206 | 24/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loteprednol Etabonate (N=206) | Vehicle (N=201)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loteprednol Etabonate (N=206) | Vehicle (N=201)
Anterior Chamber Inflammation (Eye disorders) | 7 (7) | 14 (14)
Eye Pain (Eye disorders) | 3 (3) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data generated as a result of this study will be regarded as confidential, until appropriate analysis and review by the Sponsor or its designee and the Investigator(s) are completed. The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.